CLINICAL TRIAL: NCT04195022
Title: Comparison of a Chemically Activated Composite Resin Alkasite With Resin Composite in Atypical Caries Lesions of Deciduous Teeth - A Non-inferiority Randomized Clinical Trial
Brief Title: Comparison of a Chemically Activated Composite Resin Alkasite With Resin Composite in Atypical Caries Lesions of Deciduous Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, Principal investigator, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLM2990II
Record Dates: First submitted 2019-09-30; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Deciduous teeth; Permanent dental restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemically activated Composite resin Alkasite (Experimental): Single placement of composite resin on atypical cavities.
  Interventions: Procedure: Dental Restoration with Chemically activated Composite resin Alkasite
- Bulk fill resin composite (Active Comparator): Single placement of Bulk fill resin composite on atypical cavities.
  Interventions: Procedure: Dental Restoration with Bulk fill resin composite

INTERVENTIONS:
Procedure: Dental Restoration with Chemically activated Composite resin Alkasite — Selective removal of dental caries with manual instruments, under relative isolation, application of universal adhesive system and restoration with chemically activated composite resin Alkasite.
  Arms: Chemically activated Composite resin Alkasite
Procedure: Dental Restoration with Bulk fill resin composite — Selective removal of dental caries with manual instruments, under relative isolation, application of universal adhesive system and restoration with bulk fill resin composite.
  Arms: Bulk fill resin composite

SUMMARY:
Atypical cavities, which involve more than two surfaces, one being buccal or lingual/palatal, are a challenge for restorative dentistry, since the risk of restorative failure is related to the number of surfaces involved. Thus, the purpose of this umbrella project is to conduct a randomized controlled trial (RCT) to evaluate the efficacy and patient-centered outcomes of a chemically activated composite alkasite resin in atypical deciduous molar lesions. Primary molars of children aged 4 to 7 years with at least one atypical cavitary lesion in primary molars will be selected for the RCT. The selected teeth will be randomly divided into: Alkasite chemically activated composite resin and Bulk fill composite resin. Clinical and radiographic follow-up of the lesions will be performed for 6 and 12 months. The effectiveness of the treatments will be evaluated by the longevity of the restorative procedures and paralysis of the lesions. Patient-centered outcomes will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included who have at least one posterior tooth with atypical caries lesion.

Exclusion Criteria:

* Patients with special needs will be excluded, with general health conditions that may affect the oral cavity, non-cooperating in relation to the examination, which use orthodontic apparatus and the parents/guardians or children not to consent to their participation in the study. In addition, teeth with pulp exposure, spontaneous pain, mobility, presence of swelling or fistula close to the tooth, furcation or cervical injury, teeth with restorations, sealants or enamel formation defects will be excluded.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Survival of restoration | 12 months after treatment.
  To evaluate the survival of restoration by clinical examination with FDI index.

SECONDARY OUTCOMES:
Caries lesion progression | 12 months after treatment.
  For the evaluation of caries progression, the interproximal radiographic examination will be used to verify an increase of radiolucent image under restoration.
Secondary caries lesion or on the surface adjacent to the restored tooth | 12 months after treatment.
  Presence of caries lesion on the surface adjacent to the restored tooth or on the margins of the restoration by means of visual Clinical Examination.
Perception of children and parents/guardians | 6 months after treatment.
  To evaluate the satisfaction of the children in relation to the treatment performed. The questionnaire will be used "Child's and parent's questionnaire about teeth appearance".
Operator perception | 6 months after treatment.
  It will be employed a questionnaire after the completion of the treatment performed. It will also be added a question about the behavior of children during the procedure, which will be categorized as - great behavior, regular or bad.
Parents/Guardians Satisfaction | 6 months after treatment.
  The parents/guardians will be questioned about the satisfaction regarding the treatment performed in the child. The answer will be scored by a likert scale.
Child discomfort | Immediately after the treatment.
  The child will also be questioned as to the discomfort in relation to the treatment performed. For this will be used the scale of faces of Wong-Baker.
Post Operative sensitivity of the child | 7 days after treatment.
  The child will also be questioned about the sensitivity of the restorative procedure. For this, the Wong-Baker face scale will be used.
Oral health-related quality of life | 6 months after treatment.
  The validated Brazilian version of Early Childhood Oral Health Impact Scale (ECOHIS) will be applied to children and should be answered by their parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Sao Leopoldo Mandic, Campinas, São Paulo, Brazil